CLINICAL TRIAL: NCT07275307
Title: Evaluating the Effects of Prontosan Wound Gel X on the Occurrence of Superficial Surgical Site Infections in Adult Cardiac Surgery Patients: A Single-Arm, Phase IV, Adaptive Feasibility Study
Brief Title: Impact of Prontosan Wound Gel X on Surgical Site Infections in Cardiac Surgery
Acronym: PRONTOSAN
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: B. Braun Milano SpA (Unknown)
Responsible Party: Sponsor
Other Study IDs: CET 315-2025
Record Dates: First submitted 2025-11-18; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Surgical Site Infection After Major Surgery
Keywords: Surgical site infection; SSI; Prontosan; Surgery
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Cohort: Prontosan Wound Gel X Application Group: This is a single-arm, post-marketing cohort including all adult patients (≥18 years) undergoing elective cardiac surgery via median sternotomy at IRCCS Policlinico San Donato. All enrolled participants receive the intraoperative application of Prontosan Wound Gel X, a polyhexanide-based topical antiseptic gel applied once, immediately after skin closure and before dressing placement, following a standardized, real-world surgical wound management protocol. No randomization or control group is used; all eligible patients receive the same intervention as part of routine clinical practice. The cohort is designed to evaluate the gel's effects on superficial surgical site infection occurrence, alongside secondary outcomes including length of stay, re-do surgeries, and feasibility indicators.
  Interventions: Device: Application of Prontosan Wound Gel X

INTERVENTIONS:
Device: Application of Prontosan Wound Gel X — The intervention consists of the intraoperative application of Prontosan Wound Gel X, a polyhexanide-based topical antiseptic gel, applied once immediately after skin closure and before dressing placement during elective cardiac surgery. This procedure follows a standardized surgical wound management protocol as part of routine clinical practice.

SUMMARY:
This study aims to evaluate the effects of Prontosan® Wound Gel X on the incidence of superficial surgical site infections (SSI) in adult patients undergoing elective cardiac surgery with median sternotomy. The primary objective is to assess how the intraoperative application of the gel impacts the occurrence of SSIs, defined according to CDC/NHSN criteria. Secondary objectives include evaluating the length of hospital stay, the incidence of unplanned re-operations, and identifying any latent clinical subgroups through clustering analysis.

The study will be conducted as a prospective, single-center, observational, post-market trial. The primary endpoint will be the incidence of SSIs during the post-operative hospitalization period, while secondary endpoints will focus on hospital stay duration, re-operation rates, and feasibility indicators such as adherence to the protocol and completeness of data collection. The study also includes an exploratory endpoint where hierarchical clustering will be used to identify clinical subgroups based on demographic, clinical, and procedural variables.

Up to 456 adult patients will be enrolled, all of whom are undergoing elective cardiac surgery via median sternotomy at IRCCS Policlinico San Donato. The inclusion criteria include patients aged 18 or older, scheduled for surgery, and able to provide informed consent, with the clinical decision to use Prontosan® Wound Gel X during the surgery. Exclusion criteria involve urgent surgeries, participation in other interventional studies, known hypersensitivity to the gel components, or existing skin conditions incompatible with its use.

The study duration is estimated to be approximately 18 months, depending on patient enrollment and discharge rates. The follow-up will align with the hospital stay, from the surgery date to discharge, with no post-discharge follow-up planned. Statistical analysis will include a binomial test to compare observed SSI rates with those reported in literature, while secondary data will be analyzed descriptively. An exploratory analysis will use clustering to explore latent clinical subgroups.

DETAILED DESCRIPTION:
Background Surgical site infections (SSIs) remain one of the most frequent and impactful healthcare-associated infections (HAIs) in cardiac surgery, particularly in patients undergoing median sternotomy. Despite advancements in perioperative care and infection prevention protocols, SSIs continue to pose a substantial burden on postoperative recovery, patient safety, and healthcare systems.

Superficial SSIs, which involve the skin and subcutaneous tissues, represent a significant proportion of these infections and are often underestimated in terms of their clinical implications. According to global estimates, the incidence of superficial SSIs following cardiac surgery ranges from 5% to 12%, depending on the patient population, surgical complexity, and adherence to infection control measures (Cardiothoracic Interdisciplinary Research Network et al., 2024). In Italy, recent surveillance data suggest a comparable incidence, with rates in cardiac surgery patients undergoing sternotomy reaching approximately 10-12%, particularly in high-risk groups.

The clinical consequences of superficial SSIs are far from negligible. They are associated with prolonged hospital stays, increased use of antibiotics, elevated risk of wound dehiscence, and, in some cases, progression to deeper infections such as mediastinitis. Moreover, these complications may require additional surgical interventions and intensive care, further straining healthcare resources. Economically, SSIs impose a considerable cost burden on hospitals and national health systems. Extended hospitalizations and re-operations increase direct medical costs, while indirect costs related to loss of productivity and reduced quality of life further amplify the impact. Preventing even a modest proportion of SSIs could translate into substantial cost savings and improved patient outcomes.

The development of superficial SSIs following cardiac surgery is a multifactorial phenomenon influenced by a complex interplay of intrinsic patient characteristics, procedural variables, and anatomical considerations related to the surgical approach. Intrinsic risk factors include advanced age, elevated body mass index (BMI), and the presence of comorbid conditions such as diabetes mellitus, chronic obstructive pulmonary disease (COPD), peripheral vascular disease, and immunosuppression.

These factors could compromise wound healing, increase susceptibility to infection, and impair the host immune response, thereby predisposing patients to postoperative complications, including SSIs. Procedural factors also contribute substantially to infection risk. Prolonged operative time, excessive intraoperative bleeding, use of foreign materials (e.g., sternal wires or grafts), and the overall complexity of the surgical intervention are all associated with higher rates of SSIs. Moreover, suboptimal wound management practices, including insufficient skin antisepsis or improper application of dressings, may further elevate infection risk.

Median sternotomy, the standard approach for many cardiac surgeries, presents unique challenges in SSI prevention. The anatomical location of the incision, midline, overlying the sternum, exposes it to mechanical stress from coughing, movement, or respiratory support. The surgical site is also adjacent to critical mediastinal structures, increasing the clinical severity of any infection that progresses beyond the superficial layers. Additionally, the central location of the wound increases the likelihood of contamination through hand contact or dressing manipulation during routine postoperative care.

Current SSI prevention strategies in cardiac surgery rely on a multifaceted bundle approach, integrating evidence-based measures applied throughout the perioperative continuum. These strategies aim to reduce microbial contamination, optimize host defense mechanisms, and promote proper wound healing. Intraoperative prevention protocols include the administration of prophylactic antibiotics within one hour before incision, appropriate hair removal (if necessary), strict adherence to sterile technique, and the use of antiseptic solutions such as chlorhexidine-alcohol for skin preparation. Maintaining normothermia, glycemic control, and adequate oxygenation are also recognized as critical intraoperative strategies endorsed by international guidelines, including those from the WHO and CDC. Postoperative measures focus on maintaining a clean and protected wound environment, minimizing unnecessary dressing changes, and ensuring close monitoring for early signs of infection. Patient education and staff training in wound care management also play a central role in SSI prevention.

Within this framework, topical wound care products and advanced dressings are increasingly utilized to enhance the physical barrier against microbial infiltration and to modulate the local wound environment. Antimicrobial gels, including those containing polyhexanide or other antiseptic agents, are applied directly to the surgical wound before dressing placement. These products may reduce bacterial colonization at the incision site, mitigate local inflammation, and support early tissue healing. In particular, polyhexanide-based gels offer a dual mechanism of action: antiseptic activity against a broad spectrum of pathogens and disruption of biofilm formation, which is a major contributor to chronic infection and delayed healing. When incorporated into standardized protocols, these products may complement systemic antibiotic prophylaxis and contribute to reducing superficial SSIs, especially in high-risk procedures such as cardiac surgery via sternotomy.

Although current SSI prevention protocols are comprehensive and multifactorial, superficial SSIs remain prevalent in cardiac surgery, particularly following median sternotomy. Despite the promising properties of polyhexanide-based topical agents, including broad-spectrum antimicrobial activity and biofilm disruption, their use remains largely empirical, with limited evidence from prospective, real-world studies evaluating their clinical impact. Most available data derive from heterogeneous patient populations or non-comparative case series, leaving a gap in the high-quality evidence required to support systematic integration into standard surgical care pathways. This evidence gap is especially significant given the high burden of SSIs on both patients and healthcare systems. In cardiac surgery, even superficial wound infections can lead to serious complications, including delayed recovery, reoperations, and prolonged hospitalizations, with substantial clinical and economic consequences. Given the anatomical vulnerability of sternotomy wounds and the frequency of mechanical stress in the postoperative period, targeted prophylactic strategies addressing the wound environment at the point of closure may provide critical additional protection.

Study design This is a single-cohort, post-market study employing an observational, single-arm design with adaptive stopping rules. The study is designed to evaluate the real-world effects of intraoperative application of Prontosan Wound Gel X on the occurrence of SSIs in adult patients undergoing cardiac surgery via median sternotomy. Also, the adaptive component does not involve patient-level treatment decisions but solely concerns the possibility of an early termination of enrolment once sufficient evidence on the primary endpoint has been reached.

Given the post-marketing and non-comparative nature of the study, the study does not involve randomization or a control group. Instead, all eligible patients will receive the Prontosan Wound Gel X application as part of a standardized intraoperative wound management protocol. The primary objective is to generate preliminary, real-world data on the potential benefits of Prontosan Wound Gel X in preventing superficial SSIs and to inform the design of future comparative trials.

The study adopts a flexible adaptive approach, allowing interim analyses to be conducted after every 100 patients complete their hospitalization period. These analyses will be used to: (i) evaluate early trends in SSI occurrence; (ii) assess feasibility in terms of protocol adherence and data quality; (iii) inform possible protocol modifications, including adjustments to sample size, if predefined thresholds are met. The protocol is designed to adhere to the The Adaptive designs CONSORT Extension (ACE) statement. In other words, based on these analyses, the Steering Committee will evaluate whether the pre-specified statistical threshold for the primary endpoint has already been achieved, in which case further enrolment will be discontinued to avoid exposing additional patients beyond what is ethically and scientifically necessary.

This adaptive feasibility framework allows for data-driven optimization of the study trajectory while maintaining methodological rigor. It is particularly suited to exploratory, post-marketing studies where the effect size, population heterogeneity, and operational logistics are not fully established.

The overall duration of patient participation corresponds to their entire hospital stay, from surgery to discharge, in order to capture all relevant early postoperative outcomes, including superficial SSIs, hospital length of stay, and re-do surgeries. No additional follow-up beyond discharge is planned.

Adaptive Feasibility Framework This study adopts an adaptive feasibility design, which allows for prospectively planned modifications to selected trial components based on accumulating data obtained during interim analyses. Adaptive designs are particularly suitable for exploratory, post-marketing studies where uncertainties exist regarding the effect size, population response, and operational logistics. In this context, the adaptive framework is intended to optimize the study trajectory by enabling the evaluation of early efficacy signals, assessing feasibility parameters such as protocol adherence and data quality, and informing potential refinements to the protocol, including adjustments to sample size.

Interim analyses will be conducted after every 100 patients have completed their hospitalization period. These analyses will focus primarily on the observed rate of superficial SSIs in relation to the pre-specified target threshold of 8%, as well as on the completeness and consistency of collected data and the emergence of any unexpected safety signals. Based on these interim results, the study steering committee may recommend continuation as planned, sample size recalibration, protocol modifications, or early termination of the trial. Decisions will be made in accordance with pre-specified adaptation rules designed to preserve statistical validity and scientific integrity.

The adaptation mechanism will follow a group sequential structure, with appropriate statistical safeguards, including alpha-spending functions, to control the overall type I error rate. The design is aligned with the regulatory principles outlined in the methodological and reporting standards set forth by the Adaptive Designs CONSORT Extension (ACE) statement. This approach provides both flexibility and rigor, ensuring that the study remains responsive to emerging data while maintaining transparency and reproducibility in its design and conduct.

Steering Committee

The Steering Committee will not perform any patient-level clinical or safety monitoring. Its exclusive role is to evaluate, at pre-specified interim analyses (every 100 patients), whether the primary endpoint has been reached with sufficient statistical robustness. The following rules will apply:

* Continuation of enrolment: if the observed incidence of superficial SSIs remains above the predefined threshold (≤8%) or statistical precision is not yet sufficient to draw valid conclusions.
* Early termination of enrolment: if the primary endpoint is achieved (observed incidence of superficial SSIs ≤8%) with adequate statistical power and robustness, indicating that the study objective has been met.
* Reassessment / sample size recalibration: if trends suggest a potential benefit but the level of evidence is not yet conclusive, or if data quality and completeness are insufficient to support a reliable analysis.

These decision rules are designed to ensure methodological transparency and to avoid enrolling patients beyond what is ethically necessary to address the study objectives

Prontosan Wound Gel X In this study will be recorded the use of Prontosan Wound Gel X, a polyhexanide-based topical antiseptic gel, as part of standard intraoperative wound care in cardiac surgery via median sternotomy.

This product will be applied immediately after skin closure, directly to the surgical site following cardiac surgery via median sternotomy. The application protocol is standardized and reflects real-world clinical practice: (i) after final hemostasis is achieved, sternum closed, skin sutured, and before applying the sterile dressing, a thin layer of Prontosan Wound Gel X will be spread evenly over the closed wound area using sterile technique; (ii) the surgical team will then proceed with wound dressing according to local protocol; (iii) no changes to systemic antibiotic prophylaxis or other intraoperative procedures are required as part of the study.

Overall, the product will be applied only once, during the index surgical procedure, and no repeat applications are planned. Any deviation from the standardized procedure (e.g., delayed application, use of additional topical agents) will be recorded in the case report form (eCRF) and considered in the per-protocol sensitivity analyses.

The product is CE-marked and commercially available in Europe. It will be provided by the hospital pharmacy as part of routine clinical supply, with no special labeling or randomization procedures. Its use aligns with approved indications and standard instructions for use.

Although this is a single-cohort study, all data collection will occur within a controlled hospital setting, using predefined inclusion criteria, standardized perioperative care pathways, and systematic outcomes assessment. The use of Prontosan Wound Gel X will be explicitly documented in each patient's surgical record to ensure treatment fidelity. No additional training is required for the surgical team, as the application method is simple and aligned with existing wound care practices.

Sample Size The sample size was determined based on the primary endpoint: the proportion of patients developing superficial SSIs during hospitalization. In historical cohorts of patients undergoing median sternotomy at the same institution, the incidence of superficial SSIs has ranged between 10% and 12%, which is consistent with the literature. The present study aims to detect a reduction to 8% or lower, which is considered clinically relevant in the context of real-world surgical infection prevention.

Sample size calculation was performed using G*Power (version 3.1.9.7). A one-sample binomial test (two-tailed) was used to detect a reduction in the incidence of superficial SSIs from 12% (historical reference from the context of the study, which is coherent with the literature) to 8% with the application of Prontosan Wound Gel X. A significance level (α) of 0.05 and a power of 80% were set. The required sample size was estimated to be 456 patients.

However, the study incorporates an adaptive feasibility framework with interim analyses conducted after every 100 patients. These analyses are intended to reassess the assumptions underlying the initial sample size calculation and to allow for early trial modification or termination based on observed trends. Depending on the evolving evidence regarding SSI incidence and feasibility indicators, conditional power or Bayesian posterior probabilities may be used to evaluate whether the sample size should be increased, reduced, or remain unchanged.

As this is an exploratory post-market study without a control group, no formal hypothesis testing will be applied to secondary or exploratory endpoints. The sample size is therefore driven exclusively by the primary outcome and adjusted dynamically through the adaptive design.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective cardiac surgery requiring median sternotomy (e.g., CABG, valve surgery, aortic surgery)
* Ability to provide informed consent
* Independent clinical decision by the treating surgeon to apply Prontosan Wound Gel X during surgery, irrespective of study enrollment

Exclusion Criteria:

* Urgent or emergency surgery
* Concurrent enrollment in interventional clinical trials
* Known hypersensitivity to components of Prontosan Wound Gel X
* Local skin conditions or infections at the planned incision site that preclude safe use of topical antiseptic products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (≥18 years) undergoing elective cardiac surgery via median sternotomy at IRCCS Policlinico San Donato, a high-volume cardiovascular center performing over 1,000 adult cardiac surgeries annually. Eligible participants are consecutively enrolled and represent typical real-world cardiac surgery patients undergoing procedures such as coronary artery bypass grafting, valve repair or replacement, or aortic surgery. All participants receive the intraoperative application of Prontosan Wound Gel X as part of standard wound management. The population excludes patients undergoing urgent or emergency procedures, those with contraindications to the gel, or those enrolled in interventional trials.
Sampling Method: Non-Probability Sample
Enrollment: 456 (Estimated)
Dates: Start 2026-01-08 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Superficial Surgical Site Infection (SSI) | From the day of surgery until hospital discharge, assessed for up to 30 days.
  Superficial SSIs are defined according to CDC/NHSN criteria as infections involving only the skin and subcutaneous tissue of the incision, identified by purulent drainage, positive culture from the superficial incision, or clinical signs of infection with deliberate opening by a clinician. Occurrence is assessed through daily postoperative evaluations and confirmed by an independent infectious disease specialist.

SECONDARY OUTCOMES:
Length of Hospital Stay | From the date of surgery to the date of hospital discharge, assessed for up to 30 days.
  Defined as the number of days from the date of surgery to the date of hospital discharge. Serves as an indirect marker of postoperative recovery and may reflect complications such as SSIs or delayed healing.
Incidence of Re-do Surgery | From the date of surgery until hospital discharge, assessed for up to 30 days.
  Defined as any unplanned return to the operating room for surgical re-intervention during the same hospitalization, including procedures indicated for SSI, bleeding, mechanical failure, or other clinically relevant reasons.
Protocol Adherence | From intraoperative period through postoperative hospitalization until discharge, assessed for up to 30 days.
  Proportion of surgeries in which Prontosan Wound Gel X was applied according to the standardized protocol (correct timing and technique).
Data Completeness | Assessed from the intraoperative period through discharge, for up to 30 days.
  Percentage of required study fields fully completed in the electronic case report forms.
Acceptability of Gel Use | From intraoperative period through postoperative hospitalization until discharge, for up to 30 days.
  Proportion of procedures in which the surgical team rated the intraoperative use of Prontosan Wound Gel X as acceptable.
Product-Related Adverse Events | From the day of surgery until discharge, assessed for up to 30 days.
  Incidence of adverse events considered related to Prontosan Wound Gel X, classified by type and severity.

OTHER OUTCOMES:
Identification of Latent Clinical Subgroups | From the day of surgery until hospital discharge, with analysis performed after completion of data collection; assessed for up to 30 days.
  Unsupervised hierarchical clustering (Ward's method, Euclidean distance), supported by t-SNE dimensionality reduction, will be used to identify naturally occurring patient subgroups based on demographic, clinical, and procedural variables. Cluster characteristics and associated postoperative outcomes (SSI, length of stay, re-do surgery) will be described for hypothesis generation.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Castiello, MSc, RN, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, MI, Italy

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) may be shared only upon formal request and subject to institutional review and a data use agreement. Any shared IPD will include only variables necessary for secondary analyses (e.g., demographic, clinical, procedural, and postoperative outcome data) and will exclude all direct identifiers. No individual-level data will be publicly released, and data sharing will occur solely in accordance with ethical approval and institutional policies.

REFERENCES:
- [Background] Zardi EM, Chello M, Zardi DM, Barbato R, Giacinto O, Mastroianni C, Lusini M. Nosocomial Extracardiac Infections After Cardiac Surgery. Curr Infect Dis Rep. 2022;24(11):159-171. doi: 10.1007/s11908-022-00787-0. Epub 2022 Sep 24. PMID 36187899
- [Background] Singh P, Porta A, Ranucci M, Cairo B, Gelpi F, Caruso R, Magon A, Baroni I, Conte G, Bari V. Identifying and preliminary validating patient clusters in coronary artery bypass grafting: integrating autonomic function with clinical and demographic data for personalized care. Eur J Cardiovasc Nurs. 2025 Sep 5;24(6):898-910. doi: 10.1093/eurjcn/zvaf059. PMID 40186491
- [Background] Sganga G, Baguneid M, Dohmen P, Giamarellos-Bourboulis EJ, Romanini E, Vozikis A, Eckmann C. Management of superficial and deep surgical site infection: an international multidisciplinary consensus. Updates Surg. 2021 Aug;73(4):1315-1325. doi: 10.1007/s13304-021-01029-z. Epub 2021 Mar 26. PMID 33770411
- [Background] Rosenthal VD, Yin R, Jin Z, Alkhawaja SA, Zuniga-Chavarria MA, Salgado E, El-Kholy A, Zuniga Moya JC, Patil P, Nadimpalli G, Pattabhiramarao RN, Zala D, Villegas-Mota I, Ider BE, Tumu N, Duszynska W, Nguyet LTT, Nair PK, Memish ZA. International Nosocomial Infection Control Consortium (INICC) report of health care-associated infections, data summary of 25 countries for 2014 to 2023, Surgical Site Infections Module. Am J Infect Control. 2024 Oct;52(10):1144-1151. doi: 10.1016/j.ajic.2024.04.007. Epub 2024 Apr 9. PMID 38604442
- [Background] Ragusa R, Faggian G, Rungatscher A, Cugola D, Marcon A, Mazzucco A. Use of gelatin powder added to rifamycin versus bone wax in sternal wound hemostasis after cardiac surgery. Interact Cardiovasc Thorac Surg. 2007 Feb;6(1):52-5. doi: 10.1510/icvts.2005.126250. Epub 2006 Oct 16. PMID 17669768
- [Background] Platt R, Munoz A, Stella J, VanDevanter S, Koster JK Jr. Antibiotic prophylaxis for cardiovascular surgery. Efficacy with coronary artery bypass. Ann Intern Med. 1984 Dec;101(6):770-4. doi: 10.7326/0003-4819-101-6-770. PMID 6388452
- [Background] Lee HJ, Han MY, Hwang JH, Park KJ, Shin KM, Kim ES, Lee HJ, Lim A, Han EJ, Park JY, Jang YS. Risk factors for heel pressure injury in cardiovascular intensive care unit patients. Int Wound J. 2022 Aug;19(5):1158-1164. doi: 10.1111/iwj.13711. Epub 2021 Nov 3. PMID 34734481
- [Background] Kiefer J, Harati K, Muller-Seubert W, Fischer S, Ziegler B, Behr B, Gille J, Kneser U, Lehnhardt M, Daigeler A, Dragu A. Efficacy of a Gel Containing Polihexanide and Betaine in Deep Partial and Full Thickness Burns Requiring Split-thickness Skin Grafts: A Noncomparative Clinical Study. J Burn Care Res. 2018 Aug 17;39(5):685-693. doi: 10.1093/jbcr/iry019. PMID 29668985
- [Background] Kaizer AM, Belli HM, Ma Z, Nicklawsky AG, Roberts SC, Wild J, Wogu AF, Xiao M, Sabo RT. Recent innovations in adaptive trial designs: A review of design opportunities in translational research. J Clin Transl Sci. 2023 Apr 28;7(1):e125. doi: 10.1017/cts.2023.537. eCollection 2023. PMID 37313381
- [Background] Jayakumar S, Khoynezhad A, Jahangiri M. Surgical Site Infections in Cardiac Surgery. Crit Care Clin. 2020 Oct;36(4):581-592. doi: 10.1016/j.ccc.2020.06.006. Epub 2020 Aug 12. PMID 32892815
- [Background] Hekman KE, Michel E, Blay E Jr, Helenowski IB, Hoel AW. Evidence-Based Bundled Quality Improvement Intervention for Reducing Surgical Site Infection in Lower Extremity Vascular Bypass Procedures. J Am Coll Surg. 2019 Jan;228(1):44-53. doi: 10.1016/j.jamcollsurg.2018.10.002. Epub 2018 Oct 22. PMID 30359836
- [Background] Galazzi A, Panigada M, Broggi E, Grancini A, Adamini I, Binda F, Mauri T, Pesenti A, Laquintana D, Grasselli G. Microbiological colonization of healthcare workers' mobile phones in a tertiary-level Italian intensive care unit. Intensive Crit Care Nurs. 2019 Jun;52:17-21. doi: 10.1016/j.iccn.2019.01.005. Epub 2019 Feb 5. PMID 30737099
- [Background] Downing M, Modrow M, Thompson-Brazill KA, Ledford JE, Harr CD, Williams JB. Eliminating sternal wound infections: Why every cardiac surgery program needs an I hate infections team. JTCVS Tech. 2023 Apr 14;19:93-103. doi: 10.1016/j.xjtc.2023.03.019. eCollection 2023 Jun. PMID 37324338
- [Background] De Decker I, Janssens D, De Mey K, Hoeksema H, Simaey M, De Coninck P, Verbelen J, De Pessemier A, Blondeel P, Monstrey S, Claes KE. Assessing antibacterial efficacy of a polyhexanide hydrogel versus alginate-based wound dressing in burns. J Wound Care. 2024 May 2;33(5):335-347. doi: 10.12968/jowc.2024.33.5.335. PMID 38683776
- [Background] Cooper DM, Bojke C, Ghosh P. Cost-Effectiveness of PHMB & betaine wound bed preparation compared with standard care in venous leg ulcers: A cost-utility analysis in the United Kingdom. J Tissue Viability. 2023 May;32(2):262-269. doi: 10.1016/j.jtv.2023.03.001. Epub 2023 Mar 16. PMID 36990897
- [Background] Conoscenti E, Enea G, Deschepper M, In 't Veld DH, Campanella M, Raffa G, Ragonesi B, Mularoni A, Mattina A, Blot S. A quality improvement program to reduce surgical site infections after cardiac surgery: A 10-year cohort study. Intensive Crit Care Nurs. 2025 Apr;87:103926. doi: 10.1016/j.iccn.2024.103926. Epub 2024 Dec 19. PMID 39705757
- [Background] Conoscenti E, Enea G, Deschepper M, Huis In 't Veld D, Campanella M, Raffa G, Arena G, Morsolini M, Alduino R, Tuzzolino F, Panarello G, Mularoni A, Martucci G, Mattina A, Blot S. Risk factors for surgical site infection following cardiac surgery in a region endemic for multidrug resistant organisms. Intensive Crit Care Nurs. 2024 Apr;81:103612. doi: 10.1016/j.iccn.2023.103612. Epub 2023 Dec 27. PMID 38155049
- [Background] Castiello G, Caravella G, Ghizzardi G, Conte G, Magon A, Fiorini T, Ferraris L, Devecchi S, Calorenne V, Andronache AA, Saracino A, Caruso R. Efficacy of Polyhexamethylene Biguanide in Reducing Post-Operative Infections: A Systematic Review and Meta-Analysis. Surg Infect (Larchmt). 2023 Oct;24(8):692-702. doi: 10.1089/sur.2023.199. PMID 37870810
- [Background] Cardiothoracic Interdisciplinary Research Network; Rogers LJ, Vaja R, Bleetman D, Ali JM, Rochon M, Sanders J, Tanner J, Lamagni TL, Talukder S, Quijano-Campos JC, Lai F, Loubani M, Murphy GJ. Interventions to prevent surgical site infection in adults undergoing cardiac surgery. Cochrane Database Syst Rev. 2024 Dec 2;12(12):CD013332. doi: 10.1002/14651858.CD013332.pub2. PMID 39620424
- [Background] Burnett T, Mozgunov P, Pallmann P, Villar SS, Wheeler GM, Jaki T. Adding flexibility to clinical trial designs: an example-based guide to the practical use of adaptive designs. BMC Med. 2020 Nov 19;18(1):352. doi: 10.1186/s12916-020-01808-2. PMID 33208155
- [Background] Azur MJ, Stuart EA, Frangakis C, Leaf PJ. Multiple imputation by chained equations: what is it and how does it work? Int J Methods Psychiatr Res. 2011 Mar;20(1):40-9. doi: 10.1002/mpr.329. PMID 21499542